CLINICAL TRIAL: NCT00966342
Title: Post-marketing Surveillance of Annual Influenza Vaccines: Extended Vaccine Safety and Immunogenicity Evaluation
Brief Title: Rapid Evaluation of Seasonal Influenza Vaccine
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: New studies are being offered
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. David Scheifele, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H07-01465
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Influenza
Keywords: vaccine; influenza; influenza vaccine; pandemic preparedness
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Other): Everyone gets licensed Influenza vaccine
  Interventions: Drug: Fluviral 2009/10

INTERVENTIONS:
Drug: Fluviral 2009/10 — single dose given IM .05 mL

SUMMARY:
This is an invitation to consider taking part in a research study occurring just before the upcoming influenza vaccination program across Canada. The purpose of the study is to closely assess influenza vaccine safety and immune responses, as part of a nationwide, annual surveillance project sponsored by the Public Health Agency of Canada. Such scrutiny is important given the changing nature of flu vaccines from year to year.

DETAILED DESCRIPTION:
Trivalent inactivated vaccines (TIVs) are the principal tools for minimizing seasonal influenza morbidity and mortality in populations at increased risk of adverse outcomes. To keep pace with the evolution of circulating viruses the composition of TIVs is annually updated. Depending upon circumstances, the seasonal formulation may contain 1-3 new variant strains representing Canada's supply of H1N1, H3N2 and B 2009 vaccine. Standardized manufacturing processes favour consistent vaccine safety and immunogenicity profiles from year to year but unanticipated differences can and do occur. As a consequence of the unusual occurrence of "oculorespiratory syndrome" in recipients of a Canadian-made TIV for 2000-2001, the Canadian regulatory agency has required pre-approval clinical testing of seasonal vaccines in adults. This small scale testing (120 subjects) cannot exclude the occurrence of infrequent, troublesome adverse effects. Expanded testing is desirable and would best be done soon after vaccines are approved for distribution so that results could inform the public vaccination programs that follow. Having an established capacity for rapid evaluation of a new influenza vaccine will be invaluable in the event of a pandemic, when vaccines will be less thoroughly tested before being made available to protect the public.

The objectives of this study are two-fold:

1. To assess the safety and immunogenicity of a seasonal TIV influenza vaccine quickly enough to inform subsequent public delivery programs.
2. To use the opportunity to refine preparedness for rapid evaluation of a pandemic influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

Eligibility Inclusion:

* Good general health
* Written informed consent
* Adults 20-64 years of age

Exclusion Criteria:

* compromised immune system
* allergies to eggs or thimerosol
* life-threatening reaction to previous Flu vaccine
* chronic illness, bleeding disorder

any Flu vaccine within 6 mths planning any other vaccine during study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-10 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and immunogenicity of the licensed Influenza vaccine Fluviral 2009/10 measured at 7 and 21 days for safety and 21 days for immunogenicity | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: David Scheifele, Dr., Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - KFLA Public Health Department, Kingston, Ontario
  - Mt Sinai Hospital, Toronto, Ontario
  - CHUQ de recherché, Québec, Quebec